CLINICAL TRIAL: NCT06025825
Title: Comparative Effect of Palatal Injection on Pain Perception in Pediatric Patient
Brief Title: Comparative Effect of Palatal Injection in Pediatric Patient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Kevser SANCAK, asistant professor, Ankara Yildirim Beyazıt University
Other Study IDs: 26379996/10
Record Dates: First submitted 2023-08-30; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Local Anesthetic Complication
Keywords: local anesthesia; pain
MeSH Terms: conditions — Pain | interventions — Carticaine; Epinephrine; Ultracaine D-S; Lidocaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Buccal infiltration anesthesia + palatal infiltration anesthesia (with articaine HCl): Before extraction, buccal and palatal infiltration anesthesia with articaine will perform. Following anesthesia, extraction will carry out.
  Interventions: Drug: Articaine Hydrochloride + Epinephrine
- Buccal infiltration anesthesia + palatal infiltration anesthesia (with lidocaine HCl): Before extraction, buccal and palatal infiltration anesthesia with lidocaine will perform. Following anesthesia, extraction will carry out.
  Interventions: Drug: Lidocaine Hydrochloride + Epinephrine
- Buccal infiltration anesthesia (5 minutes waiting time with articaine HCl): Before extraction, buccal infiltration anesthesia with articaine will perform. After 5 minutes, extraction will carry out.
  Interventions: Drug: Articaine Hydrochloride + Epinephrine
- Buccal infiltration anesthesia (5 minutes waiting time with lidocaine HCl): Before extraction, buccal infiltration anesthesia with lidocaine will perform. After 5 minutes, extraction will carry out.
  Interventions: Drug: Lidocaine Hydrochloride + Epinephrine
- Buccal infiltration anesthesia (8 minutes waiting time with articaine HCl): Before extraction, buccal infiltration anesthesia with articaine will perform. After 8 minutes, extraction will carry out.
  Interventions: Drug: Articaine Hydrochloride + Epinephrine
- Buccal infiltration anesthesia (8 minutes waiting time with lidocaine HCl): Before extraction, buccal infiltration anesthesia with lidocaine will perform. After 8 minutes, extraction will carry out.
  Interventions: Drug: Lidocaine Hydrochloride + Epinephrine

INTERVENTIONS:
Drug: Articaine Hydrochloride + Epinephrine — Buccal infiltration anesthesia + palatal infiltration anesthesia (with articaine HCl) was applied for first group Buccal infiltration anesthesia was applied and 5 minutes was waited before extraction.
  Buccal infiltration anesthesia was applied and 8 minutes was waited before extraction.
  Other Names: ultracaine ds
  Groups: Buccal infiltration anesthesia (5 minutes waiting time with articaine HCl); Buccal infiltration anesthesia (8 minutes waiting time with articaine HCl); Buccal infiltration anesthesia + palatal infiltration anesthesia (with articaine HCl)
Drug: Lidocaine Hydrochloride + Epinephrine — Buccal infiltration anesthesia + palatal infiltration anesthesia (with lidocaine HCl) was applied for second group Buccal infiltration anesthesia was applied and 5 minutes was waited before extraction for fourth group Buccal infiltration anesthesia was applied and 8 minutes was waited before extraction for sixth group
  Other Names: jetocaine
  Groups: Buccal infiltration anesthesia (5 minutes waiting time with lidocaine HCl); Buccal infiltration anesthesia (8 minutes waiting time with lidocaine HCl); Buccal infiltration anesthesia + palatal infiltration anesthesia (with lidocaine HCl)

SUMMARY:
The aim of this study is to compare the pain perception of pediatric patients during extraction with and without palatal injection and to show whether articaine HCl and lidocaine HCl can provide palatal anesthesia in maxillary tooth extraction without the need for a second palatal injection. In addition, to evaluate the superiority of articaine HCl and lidocaine HCl to each other in providing local anesthesia and to compare pain control between each other. An observational prospective clinical study is planned to be performed in children aged 8-12 years with maxillary tooth extraction indication. It is planned to include 96 children in the study. Patients will be divided into 6 groups. After the application of anesthesia and after tooth extraction, the pain they feel with visual analogue scale and the level of pain observed with the Wong-Baker faces pain rating scale will be marked.

DETAILED DESCRIPTION:
The study is planned to be carried out in children aged 8-12 years with maxillary tooth extraction indication. It is planned to include 96 children in the study. According to studies, under the assumption that a difference of 5 units in the number of patients would be considered significant, it was planned to include at least 5 patients in each group at 95 power and α=0.05 significance level. However, the number of patients has been updated to 96 by increasing the effect size for more meaningful results.

6 different groups will be formed in patients.

1. st group: Buccal infiltration anesthesia + palatal infiltration anesthesia (with articaine HCl)
2. nd group: Buccal infiltration anesthesia + palatal infiltration anesthesia (with lidocaine HCl)
3. rd group: Buccal infiltration anesthesia (5 minutes waiting time with articaine HCl)
4. th group: Buccal infiltration anesthesia (5 minutes waiting time with lidocaine HCl)
5. th group: Buccal infiltration anesthesia (8 minutes waiting time with articaine HCl)
6. th group: Buccal infiltration anesthesia (8 minutes waiting time with lidocaine HCl) Behavioral guidance will be given to all patients who have an indication for tooth extraction for various reasons and will be included in the study with the tell-show-do technique before treatment, after clinical and radiographic examinations. Topical anesthesia will be applied with Ultracare 20% benzocaine gel (Ultradent Products Inc., USA) for 1 minute to the mucobuccal fold area closest to the tooth to be extracted. The same application will be applied to the palatal region for the groups that will undergo palatal anesthesia. Then, for group 1, group 3 and group 5, a local anesthetic containing 1:100,000 adrenaline and articaine HCL 4%; For Group 2, Group 4 and Group 6, local anesthetic containing 20 mg/ml+0.0125 mg/ml adrenaline and lidocaine HCL was injected through a 30 gauge dental needle. 0.5 in Group 1 and Group 2. cc will be used for buccal anesthesia, 0.2 cc anesthesia will be used for palatal anaesthesia. For other groups, 1 cc of anesthesia will be administered from the buccal. After the application of local anesthesia, tooth extraction will be performed. All anesthesia applications and tooth extractions will be performed by the same pediatric dentist (E.C.T). Patients will be asked to evaluate their pain after dental anesthesia and tooth extraction separately with VAS. It will also be evaluated by the Physician performing the procedure with the Wong-Baker evaluation scale.

Among the different pain assessment methods reported in the literature, rating scales to measure their intensity are mostly used in clinical studies as they represent themselves. The VAS is one of the most commonly used self-reported measures of pain; It measures a property that is believed to change over a continuum of values that are not easy to measure directly. However, it is a one-dimensional scale that measures only the sensory component or intensity of the pain experience. The millimeter scale is the most commonly used measuring range and produces a possible score range of 0 to 100 with a 10 cm line.

The dentist who performed the tooth extraction marked the line representing the level of pain intensity perceived by the patients. The Wong-Baker faces pain rating scale (WBFPS) presents 6 faces with increasing pain rating from left to right. Each face was assigned a scale from 0 to 10 indicated on the scale... Face 0 does not hurt at all, Face 2 hurts a little, Face 4 hurts a little more, Face 6 hurts more, Face 8 hurts a lot, and Face 10 hurts as much as you can imagine' it denotes.

ELIGIBILITY:
Inclusion Criteria:

* The child has no systemic disease
* Absence of acute toothache
* Child's first tooth extraction treatment
* No suspected allergy to benzocaine, lidocaine or articaine
* Comply with Frankl's 3 or Frankl's 4 behavioral assessments

Exclusion Criteria:

* Patients who do not want to participate in the study
* Any systemic condition
* Patients with any drug or local anesthetic allergy
* Patient has acute toothache or abscess
* Patients with previous tooth extraction experience
* Frankl 1 and Frankl 2 patients

Ages: 8 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: The study is planned to be carried out in children aged 8-12 years with maxillary tooth extraction indication.
Sampling Method: Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-09-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pain during tooth extraction after anesthesia with VAS | baseline and maximum 8 minutes
  The VAS is one of the most commonly used self-reported measures of pain; It measures a property that is believed to change over a continuum of values that are not easy to measure directly. However, it is a one-dimensional scale that measures only the sensory component or intensity of the pain experience. The millimeter scale is the most commonly used measuring range and produces a possible score range of 0 to 100 with a 10 cm line
Evaluation of pain during tooth extraction after anesthesia with Wong-Baker | baseline and maximum 8 minutes
  The Wong-Baker faces pain rating scale (WBFPS) presents 6 faces with increasing pain rating from left to right. Each face was assigned a score from 0 to 10, indicated on the scale. it means that Face 0 doesn't hurt at all, Face 2 hurts a little, Face 4 hurts a little more, Face 6 hurts more, Face 8 hurts a lot, and Face 10 hurts as much as you can imagine

CONTACTS AND LOCATIONS:
Overall Officials: ceren tatlı, assist.Prof, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım beyazıt University, Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bataineh AB, Nusair YM, Al-Rahahleh RQ. Comparative study of articaine and lidocaine without palatal injection for maxillary teeth extraction. Clin Oral Investig. 2019 Aug;23(8):3239-3248. doi: 10.1007/s00784-018-2738-x. Epub 2018 Nov 12. PMID 30417227
- [Background] Raslan N, Masri R. A randomized clinical trial to compare pain levels during three types of oral anesthetic injections and the effect of Dentalvibe(R) on injection pain in children. Int J Paediatr Dent. 2018 Jan;28(1):102-110. doi: 10.1111/ipd.12313. Epub 2017 Jun 24. PMID 28646527
- [Result] Uckan S, Dayangac E, Araz K. Is permanent maxillary tooth removal without palatal injection possible? Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Dec;102(6):733-5. doi: 10.1016/j.tripleo.2005.12.005. Epub 2006 Mar 20. PMID 17138173